CLINICAL TRIAL: NCT01201200
Title: Right Ventricular Function in Patients With Obstructive Sleep Apnea Assessed by Real-time Three-dimensional Echocardiography
Brief Title: Right Ventricular Function in Patients With Obstructive Sleep Apnea
Status: Completed | Type: Observational
Sponsor: Associação Fundo de Incentivo à Pesquisa (Other)
Responsible Party: Wercules Oliveira, AFIP/Escola Paulista de Medicina
Other Study IDs: Eco2
Record Dates: First submitted 2010-09-13; First posted 2010-09-14 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2010-06

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; Right Ventricular Function; Pulmonary Hypertension
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Group 1 - Obstructive Sleep Apnea (OSA): Fifty-six patients with Obstructive Sleep Apnea
- Group 2 - Non-OSA Controls: Fifty individuals without OSA with similar age, gender and body mass index (BMI)
- Group 3 - Treatment: Fifteen patients with moderate and severe sleep apnea from group 1 underwent treatment with continuous positive airway pressure
- Group 4 - Placebo: Fifteen patients with moderate/severe sleep apnea underwent to placebo

SUMMARY:
The purpose of this study is to determine whether patients with obstructive sleep apnea have any changes in right ventricular function evaluated by three dimensional echocardiography.

DETAILED DESCRIPTION:
Several studies have reported the association between sleep disorders to an increased risk to the development of cardiac disease. However, there is no substantial that about the influence of Obstructive Sleep Apnea on the right ventricular function. Objective: to analyse the right ventricular function in patients with Obstructive Sleep Apnea by means of Real-Time Three dimensional Echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Individuals > 18 years old and < 70.

Exclusion Criteria:

* Body mass index greater than 35
* Past of clinically significant cardiac conditions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Initially, 56 patients with obstructive sleep apnea (OSA) and 50 non-OSA controls underwent real-time three-dimensional echocardiography. 30 Patients with moderate and severe OSA underwent to continuous positive airway pressure treatment over 6 months. Echocardiogram will be repeated on the third and sixth months from the treatment onset.
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2007-06; Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Orlando Campos, PhD, Study Director — Escola Paulista de Medicina
Locations (1):
- Escola Paulista de Medicina, São Paulo, São Paulo, Brazil